CLINICAL TRIAL: NCT03057093
Title: Assessment of T Wave Changes of Patients With Acute Non-ST-elevation Myocardial Infarction
Brief Title: TIII Over TI in Subjects With Myocardial Infarction
Acronym: T-infarction
Status: Completed | Type: Observational
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Dr. Fikret Er, Head of the department, University Hospital Muenster
Other Study IDs: Twave1
Record Dates: First submitted 2017-02-15; First posted 2017-02-17 (Actual); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: NSTEMI - Non-ST Segment Elevation MI
Keywords: NSTEMI, ECG
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TIII>TI: Subjects with TIII>TI in initial ECG
  Interventions: Other: Non interventional study
- Non TIII>TI: Subjects without TIII>TI in initial ECG
  Interventions: Other: Non interventional study

INTERVENTIONS:
Other: Non interventional study — retrospective noninterventional study

SUMMARY:
Study was performed to identify ECG criteria for unmasking of subjects with NSTEMI at elevated risk.

DETAILED DESCRIPTION:
In the present study the investigators assessed the value of T wave changes in subjects with NSTEMI (TIII>TI).

ELIGIBILITY:
Inclusion Criteria:

* NSTEMI and PCI

Exclusion Criteria:

* NSTEMI without percutaneous intervention

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with acute myocardial infarction without ST segment elevation
Sampling Method: Non-Probability Sample
Enrollment: 903 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2013-09-30 (Actual); Study Completion 2017-01-15 (Actual)

PRIMARY OUTCOMES:
Myocardial infarction size | 5 Days
  Assessment of myocardial damage using biomarkers

SECONDARY OUTCOMES:
Correlation with coronary artery | 1 day
  Assessment of association of infarct related artery and ECG changes

IPD SHARING:
Plan to Share IPD: No